CLINICAL TRIAL: NCT07039071
Title: Evaluation of Clinical and Patient-Reported Outcomes of Laceback: A Split-Mouth Randomised Controlled Trial
Brief Title: Evaluation of Clinical and Patient-Reported Outcomes of Laceback
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Tan Loon Han, Postgraduate Orthodontic Resident, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIUM_Laceback
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Malocclusion
Keywords: laceback; pain; plaque score; archwire; complication; breakage
MeSH Terms: conditions — Malocclusion; Pain

STUDY DESIGN:
Intervention Model Description: Split-mouth RCT - a within person trial. One side of the oral cavity will receive laceback, whereas the other side will act as control (no laceback).
Who Masked: Outcomes Assessor
Masking Description: Recording of plaque score will be blinded. Laceback and archwires will be removed, then plaque disclosing agent applied. Then plaque score will be recorded by a clinician not involved in the treatment of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laceback (Experimental): For this study, on the side of the oral cavity that is randomly allocated to receive laceback, lacebacks will be put on both upper and lower arches.
  Interventions: Device: Laceback
- No laceback (No Intervention): On the other side of the oral cavity, no laceback will be placed.

INTERVENTIONS:
Device: Laceback — Lacebacks are a kind of orthodontic auxilliaries used during the initial phase of orthodontic fixed appliance treatment, especially in premolar extraction cases. They are 0.010" stainless steel ligatures tied in figure-of-8 fashion beneath the main archwires, from the canine bracket till the first molar hook of one quadrant. For this study, on the side that is randomly allocated to receive laceback, laceback will be put on both upper and lower arches (from canine bracket to 1st molar hook).
  Arms: Laceback

SUMMARY:
The goal of this clinical trial is to evaluate oral hygiene status, archwire complications, laceback complications, and pain while using lacebacks in patients undergoing orthodontic fixed appliance treatment.

The main questions it aims to answer are:

1. What is the effect of laceback on patient's oral hygiene during alignment phase of orthodontic fixed appliance treatment?
2. What is the effect of laceback on the frequency of archwire complications during alignment phase of orthodontic fixed appliance treatment?
3. What is the frequency of laceback complications during alignment phase of orthodontic fixed appliance treatment?
4. What is the effect of laceback on pain during alignment phase of orthodontic fixed appliance treatment?

For each subject, researchers will randomly assign half of the oral cavity to receive laceback during orthodontic fixed appliance treatment, whereas the other half will not receive laceback. Researchers will then compare the effect of laceback on patient's oral hygiene, archwire complications, laceback complications, and pain.

Participants are required to carry out the usual oral hygiene practices after braces and laceback are being put up. During the observation period, they are required to notify the researcher if they suspect any breakages or loose components, so that they come to the clinic for emergency appointments. They are also required to fill up a pain diary.

DETAILED DESCRIPTION:
Aim:

To evaluate the clinical and patient-reported outcomes of laceback usage during alignment phase of orthodontic fixed appliance treatment.

Specific Objectives:

1. To assess the effect of laceback on patient's oral hygiene during alignment phase of orthodontic fixed appliance treatment.
2. To investigate the effect of laceback on the frequency of archwire complications during alignment phase of orthodontic fixed appliance treatment.
3. To determine the frequency of laceback complications during alignment phase of orthodontic fixed appliance treatment.
4. To study the effect of laceback on pain during alignment phase of orthodontic fixed appliance treatment.

Research questions:

1. What is the effect of laceback on patient's oral hygiene during alignment phase of orthodontic fixed appliance treatment?
2. What is the effect of laceback on the frequency of archwire complications during alignment phase of orthodontic fixed appliance treatment?
3. What is the frequency of laceback complications during alignment phase of orthodontic fixed appliance treatment?
4. What is the effect of laceback on pain during alignment phase of orthodontic fixed appliance treatment?

Study design:

Split-mouth randomised controlled trial. For each subject, researchers will randomly assign half of the oral cavity to receive laceback during orthodontic fixed appliance treatment, whereas the other half will not receive laceback.

Population (P) - Orthodontic patients from International Islamic University Malaysia (IIUM) aged 15 and above.

Intervention (I) - Laceback (LB) Control (C) - No laceback (no LB) Outcome (O) - Primary outcome: Plaque score (using Orthodontic Plaque Index)

Secondary outcomes:

Frequency of archwire complications Frequency of laceback complications Pain (using Visual Analogue Scale)

Study procedures:

One week after braces are put up, participants will be called back so that the researchers can put up laceback on one side of their oral cavity, and record baseline records of their oral hygiene using the Orthodontic Plaque Index (OPI). Participants are required to carry out the usual oral hygiene practices after braces and laceback are being put up. During the next three week observation period, they are required to notify the researcher if they suspect any breakages or loose components, so that they come to the clinic for emergency appointments. They are also required to fill up a pain diary for 3 weeks at specific time points, where pain will be recorded using a Visual Analogue Scale. After 3 weeks, participants will be recalled so that the researchers collect the pain diary, and record the plaque score, and any archwire/laceback complications.

Sampling method:

Convenience sampling of orthodontic patients from the Specialist and Postgraduate Orthodontic Clinic of the Kulliyyah of Dentistry, IIUM.

Sample size calculation:

Sample size is calculated based on each specific objective. Sample size calculated for specific objective 1 was the highest and was therefore chosen.

Specific objective 1 is to assess the effect of laceback on patient's oral hygiene during alignment phase of orthodontic fixed appliance treatment. A previous split-mouth study was conducted on orthodontic patients to record their plaque score using OPI. The standard deviation (SD) of OPI was calculated to be 1.88. A difference of 1 point in OPI was deemed clinically meaningful to be detected. The sample size is calculated using G*Power (Version 3.1.9.6). A total of 34 subjects are required for 68 sites (34 LB and 34 no LB), which would give a power of 85% with significance level of 0.05 to detect 1 unit difference in OPI score. Final sample size after considering 10% drop out rate is 38 patients (38 per group).

Randomisation:

Simple randomisation method will be employed. The sequence will be generated using Microsoft Excel by a co-investigator not involved in the trial. Equal number of left and right sides are allocated for laceback intervention. Sequentially numbered, opaque, sealed envelopes containing allocation card written "left" or "right" side for laceback will be prepared. As new subjects are recruited, an independent dental nurse opens the next envelope in the sequence to reveal the allocation. The prinicipal investigator is responsible for recruiting and implementing the intervention.

Blinding:

Due to the nature of the study, the participants and operator are not blinded. Some of the data collection can be blinded, i.e. recording of plaque score. During recall visits, laceback and archwires will be removed, then plaque disclosing agent will be applied. Then, plaque score will be recorded by a clinician not involved in treating the patient. All data collected will be coded and anonymised to ensure that the data analyst is blinded. The code will be held by the co-investigator and will only be revealed to the principal investigator after data analysis is completed.

Proposed statistical analysis:

Data will be analysed using IBM SPSS Statistics for Macintosh (Version 27). Normality of data will be assessed using shape of the distribution curve and Shapiro-Wilk test. Reliability assessments will be measured using Intraclass Correlation Coefficient with threshold set at 0.8 to indicate good inter- and intra-rater reliability. An intention-to-treat analysis will be employed. Missing pain scores will be imputed by last observation carried forward method.

Baseline demographic characteristics will be analysed using descriptive statistics. Plaque score, frequency of archwire complications, and pain between LB and no LB side will be compared using paired t-test or Wilcoxon signed-rank test depending on the distribution of data.

ELIGIBILITY:
Inclusion Criteria:

Patient factors

* Age 15 and above
* Medically fit and well
* Good oral hygiene - no dental caries, Basic Periodontal Examination (BPE) score 0

Orthodontic factors

* Full upper and lower arch fixed orthodontic treatment (bonded till first permanent molars)
* Pre-adjusted edgewise appliance with 0.022" slot, MBT prescription, Master Series® brackets (American Orthodontics, USA)
* Extraction of bilateral upper and lower permanent first/second premolars
* No previous orthodontic treatment

Exclusion Criteria:

* Craniofacial deformities
* Mental or physical disability leading to impaired manual dexterity, difficulty in comprehending and following oral hygiene instructions
* Underlying chronic medical illness, oral diseases

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Plaque score | T0 (baseline) - before placing laceback. T1 - 3 weeks after laceback placement.
  Plaque score will be recorded using Orthodontic Plaque Index (OPI). After removing laceback and archwires, the OPI is scored by blinded clinician after applying plaque disclosing agent on canine, premolar, first molar. Visually examine presence/absence of plaque at tooth surface adjacent to bracket base (mesial, distal, occlusal, gingival), and the condition of the gingival margin.
  The status is scored according to the criteria below:
  Score 0 - Brackets are plaque-free Score 1 - Plaque on 1 tooth surface at bracket base Score 2 - Plaque on 2 tooth surfaces at bracket base Score 3 - Plaque on 3 tooth surfaces at bracket base Score 4 - Plaque on 4 tooth surfaces at bracket base and/or gingival inflammation
  Mean OPI for LB and no LB side is calculated by adding up plaque score of all the teeth recorded on each side, and dividing it by the number of teeth scored.
  Inter and intrarater reliability testing will be done.

SECONDARY OUTCOMES:
Frequency of archwire complications | T1 - 3 weeks after laceback placement. And whenever patient comes for emergency appointment between T0 and T1.
  For the purpose of this study, archwire complications will include the following:
  * Archwire fractured at any part distal to the canine bracket - counted as one incident.
  * Archwire dislodged from one or more canine bracket, premolar bracket, or first molar tube - counted as one incident.
  * Archwire permanently deformed at any part distal to the canine bracket - counted as one incident.
  * Any combination of the above three situations - counted as one incident.
  * Whole archwire lost - counted as one incident each on both LB and no LB sides.
  Upper and lower archwires will be visually examined when the patient is first seen during the appointment. The number of complications of upper and lower archwires are summed up for each side. Total number of archwire complications throughout study period will be recorded for LB side and no LB side.
Frequency of laceback complications | T1 - 3 weeks after lacebac placement And whenever patient comes for emergency appointment between T0 and T1.
  For the purpose of this study, laceback complications will include the following:
  * Laceback ligature fractured at any part - counted as one incident.
  * Laceback ligature dislodged from one or more brackets of canine, premolar, and first molar hook - counted as one incident.
  * A combination of the above two situations - counted as one incident.
  * Whole laceback lost - counted as one incident.
  Upper and lower lacebacks will be visually examined when the patient is first seen during the appointment. The number of complications of upper and lower lacebacks are summed up. Total number of laceback complications throughout study period will be recorded. During emergency appointments, dislodged lacebacks will be retied using the same protocol described previously, whereas broken or missing laceback will be replaced using new but same type of preformed 0.010" stainless steel wire ligature (Ormco Corporation, United States of America) in the same manner.
Pain during orthodontic treatment | During appointment, T0 (baseline) - before laceback placement. Inside pain diary, between T0 to T1 at specific time points - 4 hours, 24 hours, 3 days, 1 week, 2 weeks, 3 weeks after laceback placement.
  Pain on LB and no LB side will be recorded using Visual Analogue Scale (VAS) in a pain diary. Subjects will be reminded via phone to complete the diary at home, and it will be collected back during T1. They will be asked to rate the maximum pain on each side during 4 hr, 24 hr, 3 days, 1 week, 2 weeks, 3 weeks after laceback placement. Subjects will place a mark along a 100 mm horizontal line at the most relevant position, whereby the left extreme indicates "no pain and discomfort" and the right extreme indicates "worst imaginable pain and discomfort". VAS will be measured to the nearest 1 mm using a metal ruler from the low end of the scale to the patient's mark (score 0-100). Each pain score reading will be accompanied by an open-ended question asking what is the cause of pain. Analgesics should not be taken prophylactically - score should reflect maximum pain before analgesics. From the diary, the highest pain score throughout T0-T1 is recorded for LB and no LB side.

CONTACTS AND LOCATIONS:
Overall Officials: Assistant Professor Dr. Siti Hajjar Binti Nasir, Study Chair — International Islamic University Malaysia
Locations (1):
- Department of Orthodontics, Kulliyah of Dentistry, International Islamic University Malaysia, Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Patient confidentiality. And will require permission from Director General of Health Malaysia

REFERENCES:
- [Background] Zinelis S, Eliades T, Pandis N, Eliades G, Bourauel C. Why do nickel-titanium archwires fracture intraorally? Fractographic analysis and failure mechanism of in-vivo fractured wires. Am J Orthod Dentofacial Orthop. 2007 Jul;132(1):84-9. doi: 10.1016/j.ajodo.2005.11.039. PMID 17628255
- [Background] V S B, Kaul A, Tiwari A, Aliya S, Yadav A, Bera T, Kaur Makkad P. Assessment of Various Archwire Materials and Their Impact on Orthodontic Treatment Outcomes. Cureus. 2024 Sep 18;16(9):e69667. doi: 10.7759/cureus.69667. eCollection 2024 Sep. PMID 39429425
- [Background] Usmani T, O'Brien KD, Worthington HV, Derwent S, Fox D, Harrison S, Sandler PJ, Mandall NA. A randomized clinical trial to compare the effectiveness of canine lacebacks with reference to canine tip. J Orthod. 2002 Dec;29(4):281-6; discussion 277. doi: 10.1093/ortho/29.4.281. PMID 12444268
- [Background] Sueri MY, Turk T. Effectiveness of laceback ligatures on maxillary canine retraction. Angle Orthod. 2006 Nov;76(6):1010-4. doi: 10.2319/100605-351. PMID 17090165
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Kozak U, Lasota A, Chalas R. Changes in Distribution of Dental Biofilm after Insertion of Fixed Orthodontic Appliances. J Clin Med. 2021 Nov 29;10(23):5638. doi: 10.3390/jcm10235638. PMID 34884339
- [Background] Popat H, Thomas K, Farnell DJ. Management of orthodontic emergencies in primary care - self-reported confidence of general dental practitioners. Br Dent J. 2016 Jul 8;221(1):21-4. doi: 10.1038/sj.bdj.2016.495. PMID 27388086
- [Background] Peterson BW, Tjakkes GH, Renkema AM, Manton DJ, Ren Y. The oral microbiota and periodontal health in orthodontic patients. Periodontol 2000. 2024 Jul 19. doi: 10.1111/prd.12594. Online ahead of print. PMID 39031969
- [Background] Pandis N, Walsh T, Polychronopoulou A, Katsaros C, Eliades T. Split-mouth designs in orthodontics: an overview with applications to orthodontic clinical trials. Eur J Orthod. 2013 Dec;35(6):783-9. doi: 10.1093/ejo/cjs108. Epub 2013 Feb 1. PMID 23376899
- [Background] Pandis N, Chung B, Scherer RW, Elbourne D, Altman DG. CONSORT 2010 statement: extension checklist for reporting within person randomised trials. BMJ. 2017 Jun 30;357:j2835. doi: 10.1136/bmj.j2835. PMID 28667088
- [Background] Mokhtari S, Sanati I, Babaki FA, Alamdari S, Tavana N. Investigating the effect of handedness on the dental caries pattern, gingival index, and plaque index in 6-10 years old children. Niger J Clin Pract. 2020 Apr;23(4):545-549. doi: 10.4103/njcp.njcp_600_19. PMID 32246663
- [Background] McLaughlin RP, Bennett JC. The transition from standard edgewise to preadjusted appliance systems. J Clin Orthod. 1989 Mar;23(3):142-53. No abstract available. PMID 2606968
- [Background] Marsh PD. Dental plaque as a microbial biofilm. Caries Res. 2004 May-Jun;38(3):204-11. doi: 10.1159/000077756. PMID 15153690
- [Background] Marincak Vrankova Z, Rousi M, Cvanova M, Gachova D, Ruzicka F, Hola V, Lochman J, Izakovicova Holla L, Brysova A, Borilova Linhartova P. Effect of fixed orthodontic appliances on gingival status and oral microbiota: a pilot study. BMC Oral Health. 2022 Oct 27;22(1):455. doi: 10.1186/s12903-022-02511-9. PMID 36303145
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Jiang HM, Yu C, Kan Q, Xu B, Ma C, Kang G. Effect of hydrogen on super-elastic behavior of NiTi shape memory alloy wires: Experimental observation and diffusional-mechanically coupled constitutive model. J Mech Behav Biomed Mater. 2022 Aug;132:105276. doi: 10.1016/j.jmbbm.2022.105276. Epub 2022 May 20. PMID 35642861
- [Background] Jakubovics NS, Goodman SD, Mashburn-Warren L, Stafford GP, Cieplik F. The dental plaque biofilm matrix. Periodontol 2000. 2021 Jun;86(1):32-56. doi: 10.1111/prd.12361. Epub 2021 Mar 10. PMID 33690911
- [Background] Irvine R, Power S, McDonald F. The effectiveness of laceback ligatures: a randomized controlled clinical trial. J Orthod. 2004 Dec;31(4):303-11; discussion 300. doi: 10.1179/146531204225020606. PMID 15608345
- [Background] Inauen DS, Papadopoulou AK, Eliades T, Papageorgiou SN. Pain profile during orthodontic levelling and alignment with fixed appliances reported in randomized trials: a systematic review with meta-analyses. Clin Oral Investig. 2023 May;27(5):1851-1868. doi: 10.1007/s00784-023-04931-5. Epub 2023 Mar 6. PMID 36879148
- [Background] Guzman U, Jerrold L, Abdelkarim A. An in vivo study on the incidence and location of fracture in round orthodontic archwires. J Orthod. 2013 Dec;40(4):307-12. doi: 10.1179/1465313313Y.0000000062. PMID 24297962
- [Background] Fleming PS, Johal A, Pandis N. The effectiveness of laceback ligatures during initial orthodontic alignment: a systematic review and meta-analysis. Eur J Orthod. 2013 Aug;35(4):539-46. doi: 10.1093/ejo/cjs033. Epub 2012 Apr 26. PMID 22539592
- [Background] Dowsing P, Murray A, Sandler J. Emergencies in orthodontics. Part 1: Management of general orthodontic problems as well as common problems with fixed appliances. Dent Update. 2015 Mar;42(2):131-4, 137-40. doi: 10.12968/denu.2015.42.2.131. PMID 26058226
- [Background] Beberhold K, Sachse-Kulp A, Schwestka-Polly R, Hornecker E, Ziebolz D. The Orthodontic Plaque Index: an oral hygiene index for patients with multibracket appliances. Orthodontics (Chic.). 2012;13(1):94-9. PMID 22567620
- [Background] Badran SA, Al-Zaben JM, Al-Taie LM, Tbeishi H, Al-Omiri MK. Comparing patient-centered outcomes and efficiency of space closure between nickel-titanium closed-coil springs and elastomeric power chains during orthodontic treatment. Angle Orthod. 2022 Jul 1;92(4):471-477. doi: 10.2319/120721-906. PMID 35348615
- [Background] Al-Anezi SA, Harradine NW. Quantifying plaque during orthodontic treatment: Angle Orthod. 2012 Jul;82(4):748-53. doi: 10.2319/050111-312.1. Epub 2011 Nov 1. PMID 22044115